CLINICAL TRIAL: NCT02375594
Title: Sustained Effect of a 12 Week Guided Exercise Program Conducted in an Exercise Park Equipment in the Physical Function and Physical Activity Levels of Physically Inactive Elderly: Randomized Clinical Trial
Brief Title: Exercise Park Equipment for Improving Physical Function and Physical Activity Levels in the Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacio Salut i Envelliment UAB (Other)
Collaborators: Lappset Group Oy, España (Unknown); Institut Investigacio Sanitaria Pere Virgili (Other); Atenció Primària Vallcarca - Sant Gervasi (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FSIE-LAPP-2014
Record Dates: First submitted 2015-02-09; First posted 2015-03-02 (Estimated); Last update posted 2015-03-02 (Estimated); Status verified 2015-02

CONDITIONS: Sedentary Lifestyle
MeSH Terms: conditions — Sedentary Behavior | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise in park equipment (Experimental): Participants in the intervention arm will attend a 3-month long program of 2 weekly one-hour exercise sessions in the exercise park equipment, guided by a physical therapist. The sessions will comprise a combination of aerobic, strength, balance and flexibility exercises. Up to 20 participants exercising simultaneously in the equipment under the guidance of an experienced LAPPSET physical therapist.
  Interventions: Other: Exercise in park equipment
- Control (No Intervention): Participants in the control arm will receive usual advice on healthy habits. During the study, they will be offered to attend the talks on healthy living for elderly periodically organised by their primary care centre (CAP Vallcarca - Sant Gervasi). At the end of the study, they will be invited to an exercise session at the exercise park equipment, conducted by the study physical therapist.

INTERVENTIONS:
Other: Exercise in park equipment
  Arms: Exercise in park equipment

SUMMARY:
Exercise park equipments for the elderly are designed taking into account the physical and cognitive capabilities and needs of elderly individuals. These equipments are usually built in public spaces, and may be part of public health initiatives to promote active lifestyles in the elderly.

Previous research has provided clear evidence on the short-term efficacy of exercise programs in improving physical function and level of physical activity in community-dwelling elderly. The goal of this randomized clinical trial is to assess whether an exercise intervention conducted in an exercise park equipment is able to achieve sustained improvements in physical function and level of physical activity, that are maintained for at least 3 months after the end of the intervention. The target population are community-dwelling elderly that are insufficiently active.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 70 years or more
* Insufficiently active, defined as a person who does not meet the physical activity recommendations of World Health Organization (30 minutes per day of moderate physical activity (including active leisure and travel), 5 days a week; or 30 minutes per day of vigorous physical activity, 3 days a week).

Exclusion Criteria:

* The individual refers not being able to walk 400 meters in 15 minutes or less without having to sit, lean, use a walker or require the assistance of another person.
* Moderate or severe cognitive impairment (MiniMental <19).
* Serious disease that limits physical activity (heart disease, cancer, chronic respiratory disease, joint replacements in the last 12 months, severe limitations of range of motion).
* Serious mental illness that prevents participation.
* Prescription of neuroleptic medication.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-09 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Physical performance measured with the Short Physical Performance Battery | 6 months (3 months follow up after end of intervention)
  Physical performance measured with the Short Physical Performance Battery
Amount of moderate or intense physical activity assessed with the International Physical Activity Questionnaire | 6 months (3 months follow up after end of intervention)
  Self reported weekly minutes of moderate or intense physical activity

SECONDARY OUTCOMES:
Amount of physical activity in exercise park equipment assessed with the question "Estimate in minutes the duration of any moderate or intense physical activity that you conducted last week in the exercise park equipment" | 6 months (3 months follow up after end of intervention)
  Self reported weekly minutes of moderate or intense physical activity conducted in the exercise park equipment
Fatigability measured with the Pittsburgh Fatigability Scale for Older Adults | 6 months (3 months follow up after end of intervention)
  Fatigability measured with the Pittsburgh Fatigability Scale for Older Adults
Fatigability measured with the Pittsburgh Fatigability Scale for Older Adults | 3 months (e.g. at end of intervention)
  Fatigability measured with the Pittsburgh Fatigability Scale for Older Adults
Functionality measured with the Late Life Function and Disability test | 6 months (3 months follow up after end of intervention)
  Functionality measured with the Late Life Function and Disability test
Functionality measured with the Late Life Function and Disability test | 3 months (e.g. at end of intervention)
  Functionality measured with the Late Life Function and Disability test
Social participation measured with the Index of Subjective Social Participation | 6 months (3 months follow up after end of intervention)
  Social participation measured with the Index of Subjective Social Participation
Quality of life measured with SF-12 | 6 months (3 months follow up after end of intervention)
  Quality of life measured with SF-12
Amount of moderate or intense physical activity assessed with the International Physical Activity Questionnaire | 3 months (e.g. at end of intervention)
  Weekly minutes of moderate or intense physical activity
Physical performance measured with the Short Physical Performance Battery | 3 months (e.g. at end of intervention)
  Physical performance measured with the Short Physical Performance Battery
Satisfaction assessed through open-ended questions | 3 months (e.g. at end of intervention)
  Subjective satisfaction with the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Salvà, MD, Principal Investigator — Fundació Salut i Envelliment
Locations (2):
- Spain (2):
  - CAP Vallcarca-Sant Gervasi, Barcelona
  - Fundació Salut i Envelliment, Barcelona